CLINICAL TRIAL: NCT02793466
Title: A Phase I, Open-Label, Single Institution Study to Assess the Safety, Tolerability, and Pharmacokinetics of Durvalumab in Pediatric Patients With Relapsed or Refractory Solid Tumors, Lymphoma, and Central Nervous System Tumors
Brief Title: Durvalumab in Pediatric and Adolescent Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leo Mascarenhas (Other)
Responsible Party: Sponsor-Investigator, Leo Mascarenhas, Principal Investigator, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-16-00177
Record Dates: First submitted 2016-04-22; First posted 2016-06-08 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor; Lymphoma; Central Nervous System Tumors
Keywords: Durvalumab; solid tumors; Immunotherapy; Check Point Inhibitor; pediatrics; children
MeSH Terms: conditions — Lymphoma; Central Nervous System Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab; MEDI4736 (Experimental): Open label
  Interventions: Drug: Durvalumab; MEDI4736

INTERVENTIONS:
Drug: Durvalumab; MEDI4736 — IV Infusion every 2 weeks for a maximum of 26
  Other Names: Durvalumab

SUMMARY:
This clinical trial is the first clinical trial to study Durvalumab, a checkpoint inhibitor which stimulates the patient's own immune system to act against cancer cells in children and adolescents. This trial will assess the safety and tolerability of Durvalumab in children and adolescents and also study how Durvalumab is processed in their bodies.

DETAILED DESCRIPTION:
This trial will assess the safety and tolerability of Durvalumab in children and adolescents and also study how Durvalumab is processed in their bodies.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be >12 months and <18 years of age at the time of study enrollment.
* Diagnosis: Patient must have disease that is either refractory to frontline treatment or have relapsed. Patient must have had histologic verification of a solid tumor (including lymphoma and CNS tumors) at the time of original diagnosis or relapse with the following exceptions:

  * Patients with germ cell tumors (both CNS and non-CNS) that have elevated tumor markers (e.g. α-fetoprotein, β-human chorionic gonadotropin, inhibin A/B) and radiographic evidence of disease.
  * Patients with diffuse intrinsic pontine glioma (DIPG) diagnosed by radiographic studies.
* Disease Status: Patients must have either measurable or evaluable disease that can be accurately assessed at baseline by computerized tomography (CT) or magnetic resonance imaging (MRI) and is suitable for repeated assessment with the following exception:

  * Patients with a third relapse of osteosarcoma and no measurable disease after surgical resection will be eligible for this study.
  * Therapeutic Options: Patient's current disease state must be one for which there is no known curative therapy.
* Performance Level: Karnofsky ≥ 50 for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who can actively sit up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score. See Appendix I for scoring guidelines.
* Organ Function Requirements:

  * Adequate organ and bone marrow function as defined below:
  * Absolute neutrophil count ≥ 750/mm3
  * Platelets ≥ 75,000/mm3 . Patients must be transfusion independent and should not have received a platelet transfusion within 5 days of enrollment.
  * Hemoglobin ≥8.0 g/dL. Patients may receive PRBC transfusion.
  * Adequate renal function as defined by: Creatinine clearance or radioisotope GFR > 70ml/min/m 2
  * Total serum bilirubin (conjugated plus unconjugated) ≤1.5 x upper limit of normal (ULN) for age. For patients with Hepatocellular Carcinoma (HCC) or patients with documented/suspected Gilbert's disease, bilirubin ≤3x ULN.
  * In patients with no liver metastasis: AST and ALT ≤2.5 x ULN
  * In patients with HCC or liver metastasis: AST or ALT ≤5 x ULN
  * Adequate cardiac function as indicated by shortening fraction of > 28% by echocardiogram or ejection fraction of ≥ 55% by radionuclide angiogram.
* Informed Consent: Provision of signed and dated written informed consent (parent/legal guardian if patient <18 years of age) and assent (from patients aged >7 years) prior to any study specific procedures, sampling and analyses, including screening evaluations.
* Female patients must either be of non-reproductive potential or must have a negative serum pregnancy test upon study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits as well as follow up examinations.

Exclusion Criteria:

* Prior therapy:

  * Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment.
  * Any investigational agents or study drugs from a previous clinical study within 28 days of the first dose of study treatment. Patient may be enrolled in other non-therapeutic studies.
  * Hematopoietic growth factors: Within 14 days of the last dose of a long acting growth factor (e.g. Neulasta) or within 7 days of receiving a short acting growth factor. This does not apply to erythropoetin.
  * Monoclonal antibodies: Less than 3 half-lives or 28 days (whichever is shorter) after the last dose of monoclonal antibody, and without resolution of all known toxicity of the antibody.
  * Any other chemotherapy, immunotherapy or anticancer agents within 4 weeks of the first dose of study treatment. For agents with known adverse events occurring beyond 3 weeks of administration after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * Any previous systemic exposure to a PD-1 or PD-L1 inhibitor, including Durvalumab.
  * Major surgery (excluding placement of vascular access and needle biopsies) within 2 weeks of the first dose of study treatment.
  * Radiotherapy within two weeks for local palliative XRT or within 6 weeks if craniospinal XRT or if ≥ 50% radiation of pelvis.
  * Current or prior use of immunosuppressive medication within 28 days before the first dose of Durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
  * Any prior allogeneic BMT/HSCT.
  * Autologous BMT/HSCT within 90 days.
* All prior acute toxicities from medical therapy or radiation therapy should resolve to meet the baseline inclusion criteria in regards to organ function requirement. All other prior acute toxicities that are not part of the baseline organ function requirements must improve to ≤ Grade 1 as defined in Section 5.1.1 and using CTCAE Criteria Version 4.03.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) > 470 msec obtained from at least 2 electrocardiograms (ECGs).
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block)
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Patients with hypothyroidism as a result of irradiation or thyroidectomy are also not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* Any underlying interstitial lung disease.
* Brain metastases or spinal cord compression unless asymptomatic, treated and stable for at least 1 month prior to entry into the study.
* Ongoing or expected need for systemic corticosteroids ≥10mg/day.
* Known history orf previous clinical diagnosis of tuberculosis.
* Receipt of live attenuated vaccination within 30 days prior to receiving study treatment. Inactivated viruses, such as those in the influenza vaccine, are permitted
* History of another primary malignancy within 5 years prior to starting study treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study.
* Pregnancy or Breast-Feeding: Pregnant patients are ineligible for this study due to the unknown teratogenic effects of this agent. Pregnancy tests must be obtained in females of childbearing potential prior to enrollment.
* Post-menarchal females and males who are sexually active with women of childbearing potential who are not employing/willing to employ an effective method of birth control.
* Clinically Significant Unrelated Systemic Illness: Patients with serious infections or significant pulmonary, hepatic, renal, or other end-organ dysfunction which in the judgment of the Principal or Co-Investigators would compromise the patient's ability to tolerate prescribed chemotherapy or are likely to interfere with the study procedures or results will not be eligible.
* Patient with HIV, Hepatitis B, or Hepatitis C defined by the following serology results:

  * Positive human immunodeficiency virus (HIV) antibody.
  * Positive hepatitis B surface antigen (HBsAg) and positive hepatitis B core (HBc) antibody or undetectable hepatitis B (HBV) deoxyribonucleic acid (DNA) by quantitative polymerase chain reaction (PCR) testing.
  * Positive hepatitis C (HCV) antibody or positive HCV ribonucleic acid (RNA) by quantitative PCR.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* History of hypersensitivity to Durvalumab or any excipient.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  Maximum dose of Durvalumab in milligrams per kilogram body weight that can be administered to children between the age of 1 and 18 years that will be used to study the drug further in a Phase 2 clinical trial in a population of the same age distribution
Dose Limiting Toxicity (DLT) | 28 days
  Number of patients with dose limiting toxicity
Safety Profile | Up to 15 months
  Number of patients with Adverse events
Maximum Plasma Concentration (CMax) | Up to 7 months
  Durvalumab levels micrograms/mL
Area under the curve (AUC) | 14 days
  time and Durvalumab levels days-micrograms/mL
Minimum Plasma Concentration (CTrough) | Up to 15 months
  Durvalumab levels in micrograms/mL

SECONDARY OUTCOMES:
Response rate | 8 weeks
  Objective response rate of malignancy following two cycles (4 doses) of treatment
Drug antibody level | 18 months
  Anti- Durvalumab levels in micrograms/mL
Suppression of free soluble PD-L1 suppression in serum | 15 months
  Individual soluble PDL-1 levels [pg/mL] in blood with durvalumab monotherapy
Duration of response | up to 2 years
  Time from first complete or partial response to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Leo Mascarenhas, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided